CLINICAL TRIAL: NCT01599312
Title: Forces Exerted on Upper and Lower Teeth During Intubation: a Randomized, Cross-over Trial Comparing Indirect Videolaryngoscopy to Direct Videolaryngoscopy.
Brief Title: Forces on Teeth During Videolaryngoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Catharina Ziekenhuis Eindhoven (Other)
Responsible Party: Principal Investigator, Barbe Pieters, Principal Investigator, Catharina Ziekenhuis Eindhoven
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: NL39915.060.12; M12-1217 (Other: Catharina Ziekenhuis Eindhoven)
Record Dates: First submitted 2012-05-14; First posted 2012-05-16 (Estimated); Last update posted 2015-02-10 (Estimated); Status verified 2015-02

CONDITIONS: Tooth Injuries; Intubation Complication
Keywords: Videolaryngoscopy; Forces; Teeth
MeSH Terms: conditions — Tooth Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Classic Macintosh laryngoscope (Other): Classic Macintosh laryngoscope (Karl Storz, Tuttlingen, Germany)
  Interventions: Device: Forces exerted on teeth during intubation
- McGrath® (Other): McGrath® (Aircraft Medical Ltd, Edinburgh, UK)
  Interventions: Device: Forces exerted on teeth during intubation
- C-MAC® (Other): C-MAC® (Karl Storz, Tuttlingen, Germany)
  Interventions: Device: Forces exerted on teeth during intubation
- GlideScope® Cobalt (Other): GlideScope® Cobalt (Verathon Medical, Bothell, WA, USA)
  Interventions: Device: Forces exerted on teeth during intubation

INTERVENTIONS:
Device: Forces exerted on teeth during intubation — Anesthesia will be induced in the conventional matter. The classic Macintosh laryngoscope will be placed in the patient's mouth and a tube will be brought into position in front of the glottis. Hereafter, one of the three videolaryngoscopes will be placed in the patient's mouth and the endotracheal tube will be actually passed through the vocal cords. The measurement of forces applied to the teeth will be performed using Flexiforce® sensors.
  Other Names: Macintosh laryngoscope (Karl Storz, Tuttlingen, Germany); McGrath® (Aircraft Medical Ltd, Edinburgh, UK); C-MAC® (Karl Storz, Tuttlingen, Germany); GlideScope® Cobalt (Verathon Medical, Bothell, WA, USA).; Flexiforce® sensors (A201-25, Tekscan, MA, USA)

SUMMARY:
In this randomized crossover trial the investigators test whether three different brands of videolaryngoscopes (VLS) exhibit reduced forces on both upper and lower teeth, and compare them with a classic Macintosh laryngoscope blade.

DETAILED DESCRIPTION:
During endotracheal intubation the anesthesiologist uses a laryngoscope blade to distract the tongue to achieve the best view of the glottis opening, thereby avoiding using the maxillary incisors as a fulcrum to lever the soft tissues upwards. Using the maxillary incisors as a fulcrum may otherwise result in dental trauma. It is obvious that contact with teeth and - even worse - the incidence of accidental dental trauma, is directly related to the difficulty of the intubation.

Indirect videolaryngoscopy has proven advantageous over direct laryngoscopy using a classic Macintosh blade, for improved viewing of the glottis, with subsequent more successful intubations, and a shorter effective airway time both in patients with normal and difficult airways. Previously, it has been demonstrated that the forces exerted by the anesthesiologist on the patient's maxillary incisors are reduced when using a VLS, compared with a classic Macintosh laryngoscope. However, only one type of VLS (V-MAC®, Karl Storz, Tuttlingen, Germany) was used or only forces applied to upper teeth were being registered.

ELIGIBILITY:
Inclusion Criteria:

* Informed patient consent
* ASA I -III
* Age > 18 years
* Elective surgery, other than head and/or throat surgery
* Pre-operative Mallampati I -III
* Fasted (≥6 hours)

Exclusion Criteria:

* No informed patient consent
* ASA ≥ IV
* Age < 18 year
* Emergency surgery, surgery of head and/of throat
* Locoregional anaesthesia
* Pre-operative Mallampati IV
* Fasted < 6 hours
* Pre-operative expected difficult airway
* No teeth, bad dentition
* Dental crowns and/or fixed partial denture

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-05; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Measuring the frequency with which forces are applied to the upper and lower teeth. | At intubation of the patient
  One of the three videolaryngoscopes will be placed in the patient's mouth. The measurement of forces applied to the teeth will be performed using Flexiforce® sensors.

SECONDARY OUTCOMES:
Measuring the magnitude of the forces being applied and registering the differences between (video)laryngoscopes. | At intubation of the patient

CONTACTS AND LOCATIONS:
Overall Officials: Andre A van Zundert, MD PhD FRCA, Study Director — Catharina Ziekenhuis Eindhoven
Locations (1):
- Catharina Ziekenhuis Eindhoven, Eindhoven, North Brabant, Netherlands

REFERENCES:
- [Background] Lee RA, van Zundert AA, Maassen RL, Willems RJ, Beeke LP, Schaaper JN, van Dobbelsteen J, Wieringa PA. Forces applied to the maxillary incisors during video-assisted intubation. Anesth Analg. 2009 Jan;108(1):187-91. doi: 10.1213/ane.0b013e31818d1904. PMID 19095848
- [Background] Lee RA, van Zundert AA, Maassen RL, Wieringa PA. Forces applied to the maxillary incisors by video laryngoscopes and the Macintosh laryngoscope. Acta Anaesthesiol Scand. 2012 Feb;56(2):224-9. doi: 10.1111/j.1399-6576.2011.02541.x. Epub 2011 Oct 14. PMID 22091734